CLINICAL TRIAL: NCT06573021
Title: The Role of Fluorescent Cholangiography to Improve Operative Safety in Different Severity Degree of Acute Cholecystitis During Emergency Laparoscopic Cholecystectomy.
Brief Title: Fluorescent Cholangiography in Acute Cholecystitis
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Carlo Feo, Principal investigator, University Hospital of Ferrara
Other Study IDs: 1032/2021/Oss/AUSLFe
Record Dates: First submitted 2024-08-14; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Acute Cholecystitis
Keywords: acute cholecystitis; emergency laparoscopic cholecystectomy; near-infrared fluorescent cholangiography; AAST classification
MeSH Terms: conditions — Cholecystitis, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with a clinical and radiological diagnosis of acute cholecystitis: Patients with a clinical and radiological (abdominal ultrasound and/or computed tomography) diagnosis of acute cholecystitis based on the revised Tokyo guidelines who underwent laparoscopic cholecystectomy within 24-72 hours from the onset of symptoms and patients with American Society of Anesthesiologists (ASA) score of 0-3. Near-infrared fluorescent cholangiography was performed at three time points during laparoscopic cholecystectomy: (i) following exposure of Calot's triangle, prior to any dissection; (ii) after partial dissection of Calot's triangle; (iii) after complete dissection of Calot's triangle.
  Interventions: Drug: Near-infrared fluorescent cholangiography

INTERVENTIONS:
Drug: Near-infrared fluorescent cholangiography — For intra-operative fluorescent cholangiography, 2.5 mg indocyanine green (ICG, Pulsion Medical Inc., Irving, Tx) was administered intravenously 45-60 min prior to surgery, according to the recent guidelines from the International Society for Fluorescence Guided Surgery (ISFGS) and the latest consensus conference published in 2021.

SUMMARY:
Currently, there is limited scientific evidence regarding the effectiveness of fluorescent cholangiography in emergency cholecystectomy for acute cholecystitis. The primary aim of this study was to assess the efficacy of near-infrared fluorescent cholangiography to detect extrahepatic biliary anatomy in different severity degrees of acute cholecystitis.

DETAILED DESCRIPTION:
The study aims to to evaluate the efficacy of near-infrared fluorescent cholangiography for real-time visualization of the extrahepatic biliary tree (cystic duct, common hepatic duct, cystic duct-common hepatic duct junction, common bile duct and any accessory or aberrant ducts) in emergency laparoscopic cholecystectomy before and after hepatocystic triangle dissection and in different degrees of severity of acute cholecystitis according to the American Association of Surgery for Trauma (AAST) classification, specifically distinguishing between non-gangrenous (grade I) and gangrenous or complicated (grades II-V) forms. For intra-operative fluorescent cholangiography, 2.5 mg indocyanine green (ICG) was administered intravenously 45-60 min prior to surgery, according to the recent guidelines from the International Society for Fluorescence Guided Surgery. All the operations were performed by the same team of surgeons. Near-infrared fluorescent cholangiography was performed by using Stryker's fluorescence imaging system (Stryker, Portage, Miami, USA). Near-infrared fluorescent cholangiography was performed at three defined time point during laparoscopic cholecystectomy: (i) following exposure of Calot's triangle, prior to any dissection; (ii) after partial dissection of Calot's triangle; (iii) after complete dissection of Calot's triangle, according to the "Critical View of Safety" method.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical and radiological (abdominal ultrasound and/or computed tomography) diagnosis of acute cholecystitis based on the revised TG18 who underwent laparoscopic cholecystectomy within 24-72 hours from the onset of symptoms;
* patients with ASA score of 1-3;

Exclusion Criteria:

* patients with a known allergy to indocyanine green;
* ASA score 4-5;
* patients deemed non-operable via laparoscopic approach due to high cardio-respiratory risk;
* previous surgical interventions on the biliary tract;
* history of liver cirrhosis or severe liver disease;
* ongoing pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged >18 years-old with a clinical and radiological (abdominal ultrasound and/or computed tomography) diagnosis of acute cholecystitis based on the revised Tokyo guidelines 2018 who underwent laparoscopic cholecystectomy within 24-72 hours from the onset of symptoms and patients fit for surgery with ASA score of 0-3.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of near-infrared fluorescent cholangiography in emergency cholecystectomy | From start of surgery to the end of Calot's triangle dissection
  The primary aim was to analyze the correct visualization by fluorescence of extrahepatic bile ducts (cystic duct, common hepatic duct, cystic duct-common hepatic duct junction, common bile duct, and any accessory or aberrant ducts) before and after Calot's dissection in different grades of severity of acute cholecystitis according to the AAST classification, particularly distinguishing non-gangrenous forms (grade I) from gangrenous and complicated forms (grades II-V).

SECONDARY OUTCOMES:
Conversion rate in emergency cholecystectomy by fluorescence | perioperatively
  Conversion rate (from laparoscopy to open approach)
The bail-out procedures rate in emergency cholecystectomy by fluorescence | perioperatively
  Bail-out procedures during surgery, such as subtotal cholecystectomy, antegrade cholecystectomy
The rate of bile duct injuries in emergency cholecystectomy by fluorescence | perioperatively
  Iatrogenic bile duct injuries
The duration of surgery in emergency cholecystectomy by fluorescence | perioperatively
  Total surgery duration (minutes)
Analysis of post-operative complications in emergency cholecystectomy by fluorescence | up to 30 days
  Postoperative complications according to Clavien-Dindo classification
The length of stay in emergency cholecystectomy by fluorescence | perioperatively
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: ANTONIO AP PESCE, MD PhD FACS, Study Director — Università degli Studi di Ferrara
Locations (1):
- Unità Operativa Qualità, Accreditamento, Ricerca organizzativa, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] She WH, Cheung TT, Chan MY, Chu KW, Ma KW, Tsang SHY, Dai WC, Chan ACY, Lo CM. Routine use of ICG to enhance operative safety in emergency laparoscopic cholecystectomy: a randomized controlled trial. Surg Endosc. 2022 Jun;36(6):4442-4451. doi: 10.1007/s00464-021-08795-2. Epub 2022 Feb 22. PMID 35194663
- [Background] Wang X, Teh CSC, Ishizawa T, Aoki T, Cavallucci D, Lee SY, Panganiban KM, Perini MV, Shah SR, Wang H, Xu Y, Suh KS, Kokudo N. Consensus Guidelines for the Use of Fluorescence Imaging in Hepatobiliary Surgery. Ann Surg. 2021 Jul 1;274(1):97-106. doi: 10.1097/SLA.0000000000004718. PMID 33351457
- [Background] Hernandez M, Murphy B, Aho JM, Haddad NN, Saleem H, Zeb M, Morris DS, Jenkins DH, Zielinski M. Validation of the AAST EGS acute cholecystitis grade and comparison with the Tokyo guidelines. Surgery. 2018 Apr;163(4):739-746. doi: 10.1016/j.surg.2017.10.041. Epub 2018 Jan 8. PMID 29325783
- [Background] Pesce A, La Greca G, Esposto Ultimo L, Basile A, Puleo S, Palmucci S. Effectiveness of near-infrared fluorescent cholangiography in the identification of cystic duct-common hepatic duct anatomy in comparison to magnetic resonance cholangio-pancreatography: a preliminary study. Surg Endosc. 2020 Jun;34(6):2715-2721. doi: 10.1007/s00464-019-07158-2. Epub 2019 Oct 9. PMID 31598878
- [Background] Pesce A, Piccolo G, Lecchi F, Fabbri N, Diana M, Feo CV. Fluorescent cholangiography: An up-to-date overview twelve years after the first clinical application. World J Gastroenterol. 2021 Sep 28;27(36):5989-6003. doi: 10.3748/wjg.v27.i36.5989. PMID 34629815
- [Background] Pesce A, Palmucci S, La Greca G, Puleo S. Iatrogenic bile duct injury: impact and management challenges. Clin Exp Gastroenterol. 2019 Mar 6;12:121-128. doi: 10.2147/CEG.S169492. eCollection 2019. PMID 30881079
- [Derived] Pesce A, Fabbri N, Bonazza L, Feo C. The role of fluorescent cholangiography to improve operative safety in different severity degrees of acute cholecystitis during emergency laparoscopic cholecystectomy: a prospective cohort study. Int J Surg. 2024 Dec 1;110(12):7775-7781. doi: 10.1097/JS9.0000000000002160. PMID 39806739

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/21/NCT06573021/Prot_SAP_000.pdf